CLINICAL TRIAL: NCT01409551
Title: Video-assisted Hyperthermic Pleural Chemoperfusion Versus Bed-side Talc Slurry Pleurodesis for Refractory Malignant Pleural Effusions.
Brief Title: Video-assisted Hyperthermic Pleural Chemoperfusion vs Talc Pleurodesis for Refractory Malignant Pleural Effusions.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theagenio Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Nikolaos Barbetakis, Head of Thoracic Surgery Department, Theagenio Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Theagenio Thoracic Surgery 2
Record Dates: First submitted 2011-08-03; First posted 2011-08-04 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Safety of Intervention; Efficacy of Intervention; Cost Effectiveness
Keywords: Pleural effusion; VATS; hyperthermia; thoracostomy; pleurodesis
MeSH Terms: conditions — Pleural Effusion; Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VATS hyperthermic pleural chemoperfusion (Active Comparator): The patients undergo a VATS drainage of pleural effusion with adhesiolysis and complete mobilization of the lung, following by a 1 hour hyperthermic (40oC)chemoperfusion by means of a pump machine.
  Interventions: Procedure: VATS hyperthermic chemoperfusion
- Bedside talc slurry pleurodesis (Active Comparator): The patients undergo tube thoracostomy under local anesthesia. When the lung is fully expanded, talc slurry bed-side pleurodesis is performed.
  Interventions: Procedure: Bedside talc slurry pleurodesis

INTERVENTIONS:
Procedure: VATS hyperthermic chemoperfusion — VATS, adhesiolysis, hyperthermic chemoperfusion (with a pump machine)
  Arms: VATS hyperthermic pleural chemoperfusion
Procedure: Bedside talc slurry pleurodesis — Bedside tube thoracostomy under local anesthesia. Bedside talc slurry pleurodesis.
  Arms: Bedside talc slurry pleurodesis

SUMMARY:
Aim of this study is to compare two methods of pleurodesis for refractory malignant pleural effusions, in terms of safety and efficacy.

DETAILED DESCRIPTION:
The study compares prospectively two groups of patients with refractory maignant pleural effusion. Group A consists of patients undergoing video-assisted hyperthermic pleural chemoperfusion (with a pump machine) and group B includes patients undergoing bed-side tube thoracostomy and talc slurry pleurodesis.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent symptomatic malignant pleural effusion
* No prior intrapleural therapy
* Abscence of bronchial obstruction or fibrosis preventing lung reexpansion
* No systemic chemotherapy immediately prior to or during the first 30-day interval following pleurodesis

Exclusion Criteria:

* Poor Karnofsky Performance Status

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Recurrence of pleural effusion | 2 months following intervention

SECONDARY OUTCOMES:
Morbidity | Postoperative period (7 days following intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Barbetakis, MD, PhD, Principal Investigator — Theagenio Cancer Hospital
Locations (1):
- Thoracic Surgery Department, Theagenio Cancer Hospital, Thessaloniki, Greece